CLINICAL TRIAL: NCT04008160
Title: Intelligent Underwear (IU) Monitors Pressure, Temperature, Perfusion, Humidity, and Oxygenation in Paraplegics
Brief Title: Intelligent Underwear (IU) in Paraplegics
Acronym: ProTex
Status: Withdrawn | Type: Observational
Why Stopped: responsible parties no longer available
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-04
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Skin Physiology; Spinal Cord Injuries; Pressure Injury
Keywords: perfusion; oxygenation; non invasive measurement
MeSH Terms: conditions — Spinal Cord Injuries; Pressure Ulcer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- healthy persons
  Interventions: Device: ProTex
- individuals with paraplegia
  Interventions: Device: ProTex

INTERVENTIONS:
Device: ProTex — Non invasive measurement of pressure, temperature, humidity, perfusion, and oxygenation

SUMMARY:
Pressure injuries are a major problem in patients with no or limited mobility and sensation such as paraplegics. Changes in skin physiology like changes in skin perfusion, oxygenation and humidity may explain and help to detect pressure injury development earlier. Thus, these parameters may be used for continuous monitoring of skin health. So far, there is no measuring technology available which would allow to measure continuously and quantitatively the physiological parameters, which are essential in the development of pressure injuries, over a long period of time in the clinical setting.

The goal of this pilot study is to test whether this wearable technology can be used for measurements of skin parameter and whether temperature, pressure, humidity, perfusion, and oxygenation can be measured safely and accurately.

10 healthy individuals and 10 individuals with spinal cord will be enrolled for measurements with this newly developed device over the ischium for 30 minutes. The reproducibility of the measurements will be investigated.

DETAILED DESCRIPTION:
Background of the study:

Pressure injury is a major problem in patients with no or limited mobility and sensation such as paraplegics. One of the main principles to prevent development of pressure injury is to reduce the pressure over certain regions by changing the resting or lying position periodically. Paraplegics who are suffering from loss of sensation in some parts of the body are at high risk because of the missing internal trigger to change the position regularly. Many studies have addressed the personal, social, medical and economic consequences of pressure injuries. Some studies have investigated solutions aiming to reduce the probability of pressure injury development, such as special mattresses or the frequency of moving the patients from one side to the other etc. So far it has not yet been possible to quantitatively and continuously measure the physiological skin parameters, which are essential in the development of pressure injury, over a long period of time. Up to now, long-term studies on paraplegics are limited because there are no suitable measurement devices. Current measurement devices are hard and inflexible and increase the probability of pressure ulcer development in paraplegics by applying external pressure on the tissue. In this project, the applicability of wearable measuring systems, which do not apply external pressure on the tissue, will be evaluated in paraplegics.

Aim of the study:

The goal of the study is to answer the following questions:

1. Is wearable technology usable for skin physiology measurements in paraplegics?
2. Are the measurements of skin temperature, pressure, humidity, perfusion, and oxygenation reproducible in able bodied individuals?
3. Do changes in skin temperature, pressure, humidity, perfusion, and oxygenation differ between paraplegics and healthy subjects?

Study design Two different measurement patches will be used. One patch consists of temperature, pressure, humidity and perfusion sensors. The second patch consists of near-infrared spectroscopy (NIRS) sensors (to measure oxygenation). This patch is designed for non-invasive measurement of oxygenation parameters such as oxygen saturation, oxygen consumption etc. The study is divided into two parts. The first part will be performed in 10 healthy subjects and 3 paraplegics. There will be two measurements in paraplegics and three measurements in healthy subjects, each for 10 minutes. The second part which will be conducted in 10-20 subjects (5-10 healthy and 5-10 paraplegics). The skin parameters will be measured for an hour.

Part 1a healthy subjects:

The subject will acclimatize in the room where the experiment takes place for 15 minutes. Then the patch will be placed over the ischium of the patient. Ischium will be localized manually and the patch will be placed in the underwear of the participant. The subject will be asked to sit for 10 minutes in a chair.

Part 1b paraplegics:

The subject will acclimatize in the room where the experiment takes place for 15 minutes. Then the patch will be placed over the ischium of the patient. Ischium will be localized manually and the patch will be placed in the underwear of the participant. The subject will be asked to sit for 10 minutes in a in a standard wheelchair.

Part 2:

The same procedure will be carried out with the only difference that the measurements will last 60 minutes.

Statistical Analyses:

Data will be analyzed descriptively. The reproducibility of the data will be analyzed using intraclass correlation coefficients (ICC).

The differences between data from paraplegics and that of healthy subjects will be analyzed using the Mann-Whitney-U-Test.

.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* age: 18 - 50 years

Exclusion Criteria:

* Any sign of pressure ulcer or a history of pressure ulcer on the ischium
* Diabetes
* Acute infection or disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy volunteers and individuals with paraplegia
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
change of pressure on skin | baseline and 10 minutes later
  measuring skin surface pressure with a pressure sensor in the underpants

SECONDARY OUTCOMES:
change in skin temperature | baseline and 10 minutes later
  measuring skin surface temperature with a thermometer sensor in the underpants
change in skin perfusion | baseline and 10 minutes later
  measuring skin surface perfusion with a flow sensor in the underpants
change in skin humidity | baseline and 10 minutes later
  measuring skin surface humidity with a hygrometer sensor in the underpants
change in skin oxygenation | baseline and 10 minutes later
  measuring skin oxygenation with a near-infrared spectroscopy sensor in the underpants

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Switzerland

IPD SHARING:
Plan to Share IPD: No